CLINICAL TRIAL: NCT01401335
Title: A PILOT STUDY Integrating HIV Prevention and Care With Treatment of Psychological Trauma in Vulnerable Rwandan Youth: A Community-based Pilot Intervention
Brief Title: HIV Prevention and Care of Psychological Trauma in Vulnerable Rwandan Youth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Ministry of Health, Rwanda (Other Government)
Responsible Party: Andrew R Zolopa, Stanford University School of Medicine
Allocation: Randomized | Model: Single Group | Masking: None
Other Study IDs: SU-12082010-7279; IRB# 17289 (Other: Stanford University)
Record Dates: First submitted 2011-07-19; First posted 2011-07-25 (Estimated); Last update posted 2011-07-25 (Estimated); Status verified 2011-07

CONDITIONS: Acquired Immunodeficiency Syndrome; Stress Disorders, Post-Traumatic
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Stress Disorders, Post-Traumatic | interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Trauma counseling (Other)
  Interventions: Behavioral: Questionnaires

INTERVENTIONS:
Behavioral: Questionnaires — questionnaires at entry, month 4, 8 and 12
  Other Names: trauma counseling

SUMMARY:
The investigators propose a prospective single arm pilot cohort study of 100 youth (ages 15-25) to evaluate the feasibility of this project. A convenience sample of subjects will be enrolled on a voluntary basis from those who come to the day care center located in Nyanza, a district of the Southern province, in Rwanda.

DETAILED DESCRIPTION:
The investigators propose a prospective single arm pilot cohort study of 100 youth (ages 15-25) to evaluate the feasibility of this project. A convenience sample of subjects will be enrolled on a voluntary basis from those who come to the day care center located in Nyanza, a district of the Southern province, in Rwanda. UYISENGA N'MANZI identified 400 youths in Nyanza region, organized in 4 groups, each of them between 160 to 100 youths. Many of those orphans go to school in any school in the country. This situation will be taken into account for the calendar of activities and for organization of the regular interviews and evaluations.

Random selection of the participant will be ensured by choosing study subjects from a list and attributing them an arbitrary number. The random selection will be weighted by the size of the household group across the 4 groups in the Nyanza region. Selection will also be in proportion of sex and age groups. In this manner 100 youth will be picked with 20 "backup" to account for refusals and drop-outs. Those selected youth will be asked to participate to the pilot study and will fill the consent form under the guidance of an external observer (not one of the service providers of the project to avoid consent obtained by social pressure).

Once enrolled, the subjects will be followed during 1 year with serial evaluations at baseline, 3, 6, 9 and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* 100 orphans/vulnerable youth aged 15 to 25 will be recruited through their participation at the day care center, on a voluntary basis.

Exclusion Criteria:

* Age less than 15 or greater than 25 and not participating in the day care center

Ages: 15 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 120 (Actual)
Dates: Start 2009-10; Primary Completion 2010-12 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
psychosocial interventions | 1 year
  Trauma symptoms and PTSD questionnaires.

SECONDARY OUTCOMES:
HIV treatment adherence and medical follow-up adherence questionnaires | 1 year
  HIV treatment adherence questionnaires, medical follow-up questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Andrew R Zolopa, Principal Investigator — Stanford University
Locations (2):
- Stanford University School of Medicine, Stanford, California, United States
- Uyisenga N, Kigali, KG, Rwanda